CLINICAL TRIAL: NCT03994016
Title: Preventing Adolescent Dating Violence Through Gender-Transformative Healthy Relationships Promotion: The WiseGuyz Program
Brief Title: Evaluation of the WiseGuyz Program for Adolescent Boys
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REB16-1368
Record Dates: First submitted 2019-05-10; First posted 2019-06-21 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Violence, Gender-Based
Keywords: Adolescent dating violence; Positive mental health; Sexual health

STUDY DESIGN:
Intervention Model Description: WiseGuyz' integrated and sequential curriculum is comprised of four core modules and 20 sessions per module. Sessions are a mix of targeted education, group discussion, and skills development (e.g., role play). The sequence of the modules is critical as each module builds into the next. The modules are:
  Module 1: Healthy Relationships (6 sessions) Module 2: Sexual Health (5 sessions) Module 3: Gender, Sexuality and the Media (5 sessions) Module 4: Advocacy and Leadership (4 sessions)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WiseGuyz Participant (Experimental): Individuals in this arm will receive the WiseGuyz program in their grade 9 year.
  Interventions: Behavioral: WiseGuyz
- Comparison Participant (No Intervention): Individuals in this arm will not receive any intervention in their grade 9 year, and will be used to create a matched comparison group for individuals in Arm 1 (WiseGuyz Participants).

INTERVENTIONS:
Behavioral: WiseGuyz — The WiseGuyz program was developed by the Centre for Sexuality (Calgary, AB), and aims to reduce male-perpetrated adolescent dating violence, improve mental and sexual health, and support youth to build healthier, more inclusive relationships in their peer groups, schools and communities, by helping participants identify and deconstruct gender role norms.
  WiseGuyz is offered during instructional time by community-based facilitators from the Centre for Sexuality. WiseGuyz is comprised of 20 sessions across four modules. These sessions typically take the full school year (September-May) to implement.
  Arms: WiseGuyz Participant

SUMMARY:
Adolescent dating violence (ADV) is a pressing public health problem in North America, and strategies to prevent perpetration are needed. To this end, a substantial body of research demonstrates the importance of applying a gender lens to target root causes of ADV. To date, however, there has been limited research on how to specifically engage boys in ADV prevention. As such, this protocol describes the evaluation of a program called WiseGuyz, a community-facilitated, gender-transformative healthy relationships program for mid-adolescent (~ages 13-15) male-identified youth. WiseGuyz aims to reduce male-perpetrated ADV, and improve mental and sexual health, by helping participants identify and deconstruct male gender role norms, and explore healthier, more inclusive ways of being a guy in the world. The primary goal of this evaluation is to explore the impact of WiseGuyz on ADV outcomes among mid-adolescent male-identified youth, using a mixed-methods, longitudinal, quasi-experimental design with a matched comparison group.

DETAILED DESCRIPTION:
Study Design and Overview:

In this project, the investigators will examine the association between participation in the WiseGuyz program and ADV outcomes. The investigators will use a mixed-methods, quasi-experimental design with pre-test, post-test and one-year follow-up surveys, engaging participants from two Western Canadian school divisions. Through focus groups with youth participants, the investigators will contextualize quantitative survey data, to deepen understanding of how WiseGuyz may promote the prevention of ADV.

Participants:

The investigators plan to recruit approximately 700-800 grade nine male-identified youth in 7 participating schools.

Procedures:

The investigators will make presentations on the research project to all grade 9 youth at participating schools. Any male-identified youth in grade 9 is welcome to participate, regardless of their involvement with WiseGuyz. Interested participants will need to provide signed parent/guardian consent (paper or electronic) and themselves complete an assent form to participate in the research. Quantitative data will be collected in three cohorts (Cohort One - pre-test: October 2019; post-test: May 2020; one-year follow-up: May 2021; Cohort Two - pre-test: October 2021; post-test: May 2022; one-year follow-up: May 2023; Cohort Three - pre-test: October 2022; post-test: May 2023; one-year follow-up: May 2024). An additional cohort needed to be added due to COVID-19 related study disruptions in 2019-20, 2020-21, and 2021-22.

The investigators will gather qualitative focus group data from approximately 60 WiseGuyz participants immediately post-intervention. Cohort One focus groups will occur in May 2020, Cohort Two focus groups will occur in May 2021. The investigators will also interview school leadership in Spring 2021. *note: due to COVID-19 disruptions, focus groups/interviews will only occur with Cohort 3 in Spring 2023*

To understand program implementation, implementation tracking data will be collected at the start of the program year, immediately following each WiseGuyz session, at the end of each WiseGuyz module, and at the end of the program year. The investigators will collect these data from October 2019-May 2023.

ELIGIBILITY:
Inclusion Criteria:

* all participants need to be enrolled in the 9th grade in 2019-20, 2021-22 or 2022-23 in order to participate (study length extended due to COVID-19 disruptions in 2019-20, 2020-21 and 2021-22).

Exclusion Criteria:

* individuals who are not male-identified and not in the 9th grade at one of the participating schools in 2019-20, 2021-22 or 2022-23 will not be invited to participate.

Ages: 13 Years to 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Male-identified youth (self-representation).
Enrollment: 437 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Bystander intervention behaviours for violence prevention | Cohort 1: up to 12 months; Cohort 2: up to 12 months
  Change from baseline in positive (e.g., talking to an adult) and negative (e.g., laughing) behaviours among intervention participants as compared to matched controls, as assessed using the Bystander Intervention Behaviors scale (Abebe et al., 2018).

SECONDARY OUTCOMES:
Adolescent dating violence perpetration | Cohort 1: 12 months; Cohort 2: 12 months
  Change from baseline in overall perpetration (physical, sexual and/or psychological) among intervention participants as compared to matched controls, as assessed using the Conflict In Adolescent Dating Relationships Inventory (CADRI; Wolfe et al., 2001).
Positive mental health | Cohort 1: 12 months; Cohort 2: 12 months
  Change from baseline in overall positive mental health (emotional, social and psychological) among intervention participants as compared to matched controls, as assessed using the Mental Health Continuum-Short Form (MHC-SF; Keyes, 2006).
Bullying perpetration | Cohort 1: 12 months; Cohort 2: 12 months
  Change from baseline in overall bullying perpetration (physical, verbal, social, cyber) among intervention participants as compared to matched controls, as assessed using the School Climate Bullying Survey - Bullying Behavior Sub-Scale (SCBS-BB; Cornell, 2016).
Friendship closeness | Cohort 1: 12 months; Cohort 2: 12 months
  Change from baseline in overall friendship closeness (emotional support, intimate disclosure, companionship, approval, satisfaction) among intervention participants as compared to matched controls, as assessed using the Network of Relationships Inventory - Relationship Qualities Version (NRI-RQV; Buhrmester & Furman, 2008).
Homophobic name-calling | Cohort 1: 12 months; Cohort 2: 12 months
  Change from baseline in homophobic name-calling among intervention participants as compared to matched controls, as assessed using the Homophobic Content Agent Scale (Poteat & Espelage, 2007).
Sexual health self-efficacy | Cohort 1: up to 12 months; Cohort 2: up to 12 months
  Change from baseline in sexual health self-efficacy among intervention participants as compared to matched controls, as assessed using the Sexual Health Self-Efficacy Scale (Barthalow et al., 2010).
Adherence to male role norms | Cohort 1: Immediate post-test; Cohort 2: Immediate post-test
  Change from baseline in adherence to male role norms promoting emotional restriction, avoidance of femininity and toughness among intervention participants as compared to matched controls, as assessed using the Male Role Norms Inventory-Adolescent-Revised (MRNI-A-r; Levant et al., 2012).
Attitudes towards sexual minorities | Cohort 1: Immediate post-test; Cohort 2: immediate post-test
  Change from baseline in negative attitudes towards sexual minorities among intervention participants as compared to matched controls, as assessed using the Negativity Towards Sexual Minorities scale (NTSM; Levant et al., 2012).
Dating abuse awareness | Cohort 1: Immediate post-test; Cohort 2: Immediate post-test
  Change from baseline in dating abuse awareness among intervention participants as compared to matched controls, as assessed using the Dating Abuse Awareness Scale (Abebe et al., 2018).
Intentions to intervene with peers | Cohort 1: Immediate post-test; Cohort 2: Immediate post-test
  Change from baseline in intentions to intervene with peers (positive bystander behaviour for violence prevention) among intervention participants as compared to matched controls, as assessed using the Intentions to Intervene with Peers scale (Abebe et al., 2018).
Help-seeking | Cohort 1: Immediate post-test; Cohort 2: Immediate post-test
  Change from baseline in intentions to seek help for behavioural health problems among intervention participants as compared to matched controls, as assessed using the General Help-Seeking Questionnaire (GHSQ; Wilson et al., 2005).

CONTACTS AND LOCATIONS:
Overall Officials: Deinera Exner-Cortens, PhD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data from this project may be preserved in a publicly accessible, secure and curated repository or other platform for discovery and reuse by others, but these data will not allow for any identification of individual participants. The investigators are still preparing our IPD sharing plan, and will upload once it is finalized.
Supporting Information: Study Protocol, ICF
Time Frame: Within three years of completion of study

REFERENCES:
- [Background] Exner-Cortens D, Hurlock D, Wright A, Carter R, Krause, P. Preliminary evaluation of a gender-transformative healthy relationships program for adolescent boys [published online ahead of print January 31, 2019]. Psychol Men Masculin. doi:10.1037/men0000204
- [Background] Claussen C. Men engaging boys in healthy masculinity through school-based sexual health education [published online ahead of print August 10, 2018]. Sex Education. doi:10.1080/14681811.2018.1506914
- [Background] Claussen C. The WiseGuyz Program: Sexual health education as a pathway to supporting changes in endorsement of traditional masculinity ideologies. The Journal of Men's Studies. 25(2): 150-167, 2016.
- See also: Information on the WiseGuyz program — https://www.centreforsexuality.ca/programs-workshops/wiseguyz/